CLINICAL TRIAL: NCT06740500
Title: Effect of Bifidobacterium Animalis Subsp. Lactis Bi66 Supplementation on Gut Function in Healthy Adults: a Double-blind Randomized Controlled Trial
Brief Title: Effect of Bifidobacterium Animalis Subsp. Lactis Bi66 Supplementation on Gut Function in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YY202411
Record Dates: First submitted 2024-12-15; First posted 2024-12-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy Adult
Keywords: probiotic; Bifidobacterium animalis subsp. lactis Bi66; bowel movement frequency; gut microbiota
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic Bi66 (Experimental): Bi66 group adminster a sachet of probiotic powder (1 g), including Bifidobacterium animalis subsp. lactis Bi66 6.0 × 1010 CFU and a maltodextrin carrier once daily for 8 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo group adminster a sachet of placebo powder (1 g) containing maltodextrin once daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — probiotic sachet mainly contains Bifidobacterium animalis subsp. lactis Bi66 and maltodextrin.
  Other Names: Bifidobacterium animalis subsp. lactis Bi66
  Arms: Probiotic Bi66
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn the effect of Bifidobacterium animalis subsp. lactis Bi66 supplementation on gut function in healthy adults. The main questions it aims to answer are:

1. Does Bi66 affect the gut function(bowel movement frequency and stool form)?
2. Does Bi66 affect the gut microbiota and short-chain fatty acids ? Researchers will compare probiotic Bi66 to a placebo (a look-alike substance that contains no Bi66) to see if Bi66 works to affect gut function.

Participants will

1. Take Bi66 or a placebo every day for 8 months
2. Return the used sachets and stool diaries every 7 days and record bowel movement frequency per week and Bristol Stool Scale
3. Have checkups, including questionnaire survey, physical measurement, dietary survey, collection and detection of biological samples at baseline, week 4, week 8

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* Self-reported bowel movement frequency less than 5 times per week;
* Change of weight no more than 3 kg within the last 2 months；
* No consumption of probiotics, prebiotics, synbiotics within the last 2 months

Exclusion Criteria:

* Pregnant or breastfeeding women；
* Smoking；
* BMI < 18 kg/m2 or ≥28 kg/m2；
* Suffering from gastrointestinal disorders such as gastroenteritis, gastroduodenal ulcer, ulcerative colitis, Crohn's disease, intestinal stress syndrome, functional diarrhea, gastroparesis, etc；
* History of gastrointestinal surgery (except appendectomy or hernia repair)；
* Change in dietary habits within the last 1 month (e.g. ketogenic diet, etc.)；
* History of major surgery within the last 3 months or major surgery planned in the next 1 month;
* Use of antibiotics, acid-suppressing drugs, pro-digestive drugs (gastrointestinal, morpholine, cisapride, etc.), anti-constipation drugs, anti- diarrhea drugs, etc., in the last 1 month;
* Participate in a similar intervention study within the last 1 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Bowel movement frequency | From enrollment to the end of supplementation at 8 weeks
  Bowel movement frequency per week will be measured by stool diary
gut microbiota | Baseline, 4 weeks, 8 weeks
  The fecal microbiota will be measured using 16S rRNA gene amplicon sequencing and change in the composition of beneficial bacteria will be measured using Quantitative Real-time polymerase chain reaction.

SECONDARY OUTCOMES:
Stool form | From enrollment to the end of supplementation at 8 weeks
  stool form will be measured by the Bristol Stool Scale (BSS)
Fecal short-chain fatty acids | Baseline, 4 weeks, 8 weeks
  Fecal short-chain fatty acids will be measured by gas chromatography-mass spectrometry (GC-MS)
Inflammatory cytokine | Baseline, 4 weeks, 8 weeks
  Fasting plasma inflammatory cytokine, including CRP, IL-1β, IL-6, IL-8, IL-10, TNF-α, and IFN-γ will be measured by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Liegang Liu, PhD, Principal Investigator — School of Public Health, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No